CLINICAL TRIAL: NCT03647267
Title: Randomized Clinical Trial Assessing the Effects of Pneumatic Vitreolysis on Vitreomacular Traction
Brief Title: Effects of Pneumatic Vitreolysis on Vitreomacular Traction
Acronym: AG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRCR.net Protocol AG; U10EY014231 (NIH); U10EY023207 (NIH)
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Vitreomacular Traction
MeSH Terms: interventions — Observation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Visual acuity and optical coherence tomography technicians will be masked to treatment group at all visits. The goal is for study participants to remain masked to their treatment group assignment, although it is likely that the gas bubble will be visible to participants in the pneumatic vitreolysis group. Investigators and study coordinators are not masked to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pneumatic Vitreolysis (Active Comparator): Participants randomized to the Pneumatic Vitreolysis arm will receive 0.3-mL intraocular injection of C3F8 gas.
  Interventions: Device: Pneumatic Vitreolysis (C3F8 injection)
- Observation (Placebo Comparator): Participants randomized to the observation group will receive a sham injection.
  Interventions: Other: Observation

INTERVENTIONS:
Device: Pneumatic Vitreolysis (C3F8 injection) — Pneumatic Vitreolysis will be performed via an intraocular injection of C3F8 gas. Perfluoropropane (C3F8) is an inert gas under pressure and is administered by injection into the vitreous cavity. It was approved by the FDA in February 1993 (P900066) for the use of placing pressure on detached retina.
  Arms: Pneumatic Vitreolysis
Other: Observation — No intervention; sham injection only
  Arms: Observation

SUMMARY:
Eyes with idiopathic symptomatic vitreomacular traction (VMT) without a macular hole will be randomly assigned to 0.3-mL intraocular gas (C3F8) injection or sham injection to determine if pneumatic vitreolysis (PVL) is effective in releasing VMT.

DETAILED DESCRIPTION:
Investigational Device: 0.3-mL intraocular gas (C3F8) injection

Objectives

Primary

1. To compare the proportion of eyes with central VMT release on OCT after pneumatic vitreolysis with gas injection versus observation (sham injection) in eyes with VMT without an associated macular hole.

   Secondary
2. To evaluate visual function outcomes at 24 weeks after gas injection is performed compared with sham injection.

Study Design: Multi-center, randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. At least one eye meets the study eye criteria listed below.
2. Able and willing to provide informed consent.
3. Able and willing to avoid high altitude travel, including airline travel, until gas resolution (approximately 6 to 8 weeks).
4. For phakic patients, able and willing to avoid supine position until gas resolution (approximately 6 to 8 weeks).
5. Able and willing to wear wristband that informs any medical personnel that the patient has a gas bubble in the eye

   Exclusion

   A potential participant is not eligible if any of the following exclusion criteria are present:
6. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status that might preclude completion of follow-up)
7. Participation in an investigational trial within 30 days of randomization that involves treatment with any drug or device that has not received regulatory approval for the indication being studied at the time of study entry

   • Note: study participants should not receive another investigational drug/device while participating in the study
8. Known contraindication to any component of the treatment
9. Known allergy to any drug used in the procedure prep (including povidone iodine)
10. Potential participant is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next 6 months following randomization
11. Anticipated surgery requiring anesthesia within the next 6 months following randomization

    • Participants cannot receive nitrous oxide until gas resolution
12. For women of child-bearing potential, pregnant at the time of enrollment

    • Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgement may be used to determine when a pregnancy test is needed.

    Study Eye Criteria

    The participant must have at least one eye meeting all of the inclusion criteria and none of the exclusion criteria listed below.

    A participant can have only one study eye. If both eyes are eligible at the time of randomization, the study eye will be selected by the investigator and participant before randomization.

    The eligibility criteria for a study eye are as follows:

    Inclusion
    1. Vitreomacular adhesion on OCT that is no larger than 3000 microns with visible separation of the vitreous on either side as seen on horizontal and vertical scans, confirmed by central reading center Note: presence of epiretinal membrane is neither a requirement nor exclusion.
    2. Decreased visual function (e.g. metamorphopsia or other visual symptom) that is attributed to VMT.

    Examples of visual symptoms include:

    a) Distortion and/or reduction in visual acuity b) Recognized difficulty with reading, driving, or using a computer c) Patient recognized interference with quality of life because of a and/or b.

    c. Visual acuity letter score of at least 19 (approximate Snellen equivalent 20/400 or better) and at most 78 (20/32 or worse) d. Investigator and participant willing to wait 6 months before surgical intervention, provided visual acuity remains stable

    • An eye that requires prompt treatment for VMT should not be enrolled

    Exclusion e. Other ocular condition that might affect visual acuity during the course of the study or require intraocular treatment (e.g., retinal vein occlusion, substantial age-related macular degeneration, or macular edema induced by a condition other than VMT) • If diabetic retinopathy is present, severity level must be microaneurysms only or better (≤ diabetic retinopathy severity level 20)

    • Presence of drusen is acceptable; however, eyes with geographic atrophy or neovascular age-related macular degeneration involving the macula are excluded f. High level of myopia (spherical equivalent of -8.00 diopters or more myopic if phakic or retinal abnormalities consistent with pathologic myopia if phakic or pseudophakic) g. History of prior gas injection, ocriplasmin injection, or intraocular injection for any reason h. History of prior vitrectomy i. History of uncontrolled glaucoma

    • IOP must be <30 mmHg, with no more than one topical glaucoma medication, and no documented glaucomatous field loss for the eye to be eligible j. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or major ocular surgery anticipated within the next 6 months following randomization k. History of YAG capsulotomy performed within 4 months prior to randomization l. Aphakia or anterior chamber intraocular lens m. Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis n. Uveitis o. Presence of any macular hole or lamellar hole (according to reading center grading) p. Retinal history or pathology that might predispose an eye to an increased risk of retinal detachment from the procedure

    • Untreated retinal tears, not retinal holes, are an exclusion. It is up to the investigator to determine whether extent of lattice degeneration or other pathology might increase the risk of retinal detachment.

    q. Any contraindication to paracentesis (e.g., history of narrow angle glaucoma) r. Lenticular or zonular instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clement Chan, MD, Study Chair — Southern California Desert Retina Consultants, MC
Locations (41):
- United States (41):
  - Retinal Diagnostic Center, Campbell, California
  - Atlantis Eye Care, Huntington Beach, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - East Bay Retina Consultants, Inc, Oakland, California
  - Southern California Desert Retina Consultants, MC, Palm Desert, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida College of Med., Dept of Ophthalmology, Jacksonville Hlth Sci Ctr, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Retina Institute, Orlando, Florida
  - Southeast Eye Institute, PA dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Gailey Eye Clinic, Bloomington, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Illinois Retina Associates, S.C., Oak Park, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Mid-America Retina Consultants, P.A., Overland Park, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - Elman Retina Group, PA, Baltimore, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Mayo Clinic Department of Opthalmology, Rochester, Minnesota
  - The Retina Institute, St Louis, Missouri
  - MaculaCare, New York, New York
  - Western Carolina Clinical Research, LLC, Asheville, North Carolina
  - Charlotte Eye, Ear, Nose, and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc, Beachwood, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Oregon Retina, LLP, Eugene, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Spokane Eye Clinic, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Pneumatic Vitreolysis (PVL): Pneumatic vitreolysis is an in-office intraocular injection of an expansile gas (C3F8) to induce release of vitreomacular traction.
- Sham: For sham injections, the hub of a needleless syringe was pressed against the conjunctival surface to simulate the pressure of an injection.
Period: Overall Study
Arm/Group | Pneumatic Vitreolysis (PVL) | Sham
Started | 24; 24 Eyes | 22; 22 Eyes
Completed | 23; 23 Eyes | 22; 22 Eyes
Not Completed | 1; 1 Eyes | 0; 0 Eyes
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumatic Vitreolysis (PVL) | Sham | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (10) | 75 (8) | 72 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 16 | 17 | 33
  Hispanic or Latino | 4 | 5 | 9
  non-Hispanic Black/African American | 3 | 0 | 3
  Unknown or not reported | 1 | 0 | 1
Diabetes Type [Count of Participants; unit: Participants]
  No | 16 | 12 | 28
  Type 2 | 8 | 10 | 18
E-ETDRS visual acuity letter score [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
  units on a scale | 67.8 (10.3) | 69.2 (8.4) | 68.5 (9.4)
Intraocular pressure [Mean (Standard Deviation); unit: mmHg] | 15 (4) | 14 (3) | 15 (4)
Lens status on clinical exam [Number; unit: Eyes]
  Phakic (natural lens) | 14 | 9 | 23
  Posterior Chamber intraocular lens | 10 | 13 | 23
Epiretinal membrane in central subfield [Number; unit: Eyes] — Randomization stratification factor
  Eyes | 2 | 1 | 3
Width of vitreomacular attachment that extends within the central subfield [Median (Inter-Quartile Range); unit: Microns] | 480 [315 to 694] | 503 [427 to 646] | 495 [342 to 682]
Loss of ellipsoid zone integrity in central subfield [Number; unit: Eyes] | 15 | 8 | 23
Loss of ellipsoid zone integrity in foveal center [Number; unit: Eyes] | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Central Vitreomacular Traction Release Without Rescue Vitrectomy
Time Frame: at 24 Weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL) | Sham
Number analyzed (Participants) | 23 | 22
Number analyzed (Eyes) | 23 | 22
percentage of eyes | 78 | 9

2. Secondary Outcome: Number of Eyes With Rescue Treatment Before the 24-week Visit
Time Frame: up to 24 weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL) | Sham
Number analyzed (Participants) | 23 | 22
Number analyzed (Eyes) | 23 | 22
Eyes | 1 | 0

3. Secondary Outcome: Number of Eyes With Rescue Vitrectomy Completed Before the 24-week Visit or Planned at the 24 Week Visit
Description: scheduled rescue vitrectomy must be completed within the subsequent 12 weeks.
Time Frame: through 24 Weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis | Observation
Number analyzed (Participants) | 23 | 22
Number analyzed (Eyes) | 23 | 22
Eyes | 1 | 1

4. Secondary Outcome: Number of Eyes With Central Vitreomacular Traction Status
Time Frame: up to 24 weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis | Observation
Number analyzed (Participants) | 23 | 22
Number analyzed (Eyes) | 23 | 22
Eyes
  Released without rescue vitrectomy | 18 | 2
  Released with rescue vitrectomy | 1 | 0
  Not released and no rescue vitrectomy | 4 | 20
  Not released despite rescue vitrectomy | 0 | 0

5. Secondary Outcome: Mean Change in E-ETDRS Visual Acuity Letter Score From Baseline
Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis | Observation
Number analyzed (Participants) | 23 | 22
Number analyzed (Eyes) | 23 | 22
units on a scale | 6.7 (12.4) | 6.1 (9.6)

6. Secondary Outcome: Mean Change in E-ETDRS Visual Acuity Letter Score From Baseline
Description: as for outcome 5
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis | Observation
Number analyzed (Participants) | 23 | 22
Number analyzed (Eyes) | 23 | 22
units on a scale | 6.7 (12.4) | 6.1 (9.6)

ADVERSE EVENTS:
Time Frame: 24- weeks
Arm/Group | Pneumatic Vitreolysis | Observation
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 5/24 | 0/22
Other Adverse Events (participants affected / at risk) | 10/24 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumatic Vitreolysis (N=24) | Observation (N=22)
Cataract traumatic (ocular injury) (Eye disorders) | 1 (1) | 0 (0)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 2 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumatic Vitreolysis (N=24) | Observation (N=22)
Anterior chamber cell (Eye disorders) | 1 (1) | 0 (0)
Anterior chamber flare (Eye disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Conjunctival hyperemia (Eye disorders) | 0 (0) | 1 (1)
Corneal abrasion (Eye disorders) | 0 (0) | 1 (1)
Corneal edema (Eye disorders) | 1 (1) | 0 (0)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0)
Eye itching (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Nuclear sclerosis (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 2 (2) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0)
Posterior vitreous detachment (Eye disorders) | 3 (3) | 0 (0)
Stye (Eye disorders) | 0 (0) | 1 (1)
Subconjunctival hemorrhage (Eye disorders) | 2 (2) | 0 (0)
Visual disturbances (Eye disorders) | 1 (1) | 0 (0)
Visual flashes (Eye disorders) | 0 (0) | 1 (1)
Vitreous debris (Eye disorders) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03647267/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03647267/SAP_001.pdf
  • Informed Consent Form (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03647267/ICF_002.pdf